CLINICAL TRIAL: NCT01606774
Title: A Modernized Approach to Prenatal Care in Low Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Allan Nadel, Director of Prenatal Diagnosis, Dept. of OB/GYN, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNC2.0
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Pre-eclampsia; Intrauterine Growth Retardation
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low risk patients (Experimental): Patients who agreed to 4 telemedicine obstetrical visits
  Interventions: Other: Modernized prenatal care

INTERVENTIONS:
Other: Modernized prenatal care — Home monitoring/phone surveillance/28 week ultrasound in place of 4-5 routine prenatal visits between 18 and 36 weeks

SUMMARY:
The investigators plan to identify 80 pregnant women at low risk for obstetrical complications and replace 4-5 routine third trimester visits with a structured program of home weight, blood pressure and urine protein monitoring along with regular structured phone interviews and a 28 week ultrasound. The investigators hypothesis is that this protocol is both safe and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Age < 35
* Doesn't live alone
* Current phone number
* Previous pregnancy
* No prior second trimester miscarriage/fetal loss after 13 weeks
* Previous delivery
* If yes, all had uncomplicated antepartum course
* All Deliveries > 37 weeks
* All birth weight > 2700 grams
* Maternal BMI between 18.5 and 30
* No chronic medical problems
* No current substance abuse
* Spontaneous conception
* No family history of pre-eclampsia
* Agrees to first trimester aneuploidy screening

Exclusion Criteria:

* Clinically significant abnormalities on routine physical exam or routine laboratory results
* Multiple pregnancy
* Fetal abnormalities detected on either the 11-14 week or the 18 week ultrasound including a nuchal translucency > 3 mm but not including second trimester markers for aneuploidy or a low lying placenta
* A risk of fetal aneuploidy on first trimester screening > 1:300 PAPP-A < 5 %ile or HCG < 1 %ile (abnormalities of these serum analytes routinely obtained as part of aneuploidy screening are associated with an increased risk of adverse outcome)
* Elevated blood pressure (> 140/90),
* Cervical length < 3 cm at the 18 week ultrasound (which is associated with an increased risk for preterm delivery).

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Unanticipated pregnancy complications | Gestational age 18-36 weeks
  Any maternal and/or fetal adverse outcome that was not detected, but could have been detected by routine antepartum visits between 18 and 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Nadel, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicolaides KH. A model for a new pyramid of prenatal care based on the 11 to 13 weeks' assessment. Prenat Diagn. 2011 Jan;31(1):3-6. doi: 10.1002/pd.2685. No abstract available. PMID 21210474